CLINICAL TRIAL: NCT01782092
Title: Effect of Activator Methods Technique on Lowering A1c Levels in Type II Diabetics
Brief Title: Activator and Type II Diabetics
Status: Completed | Type: Observational
Sponsor: Life University (Other)
Responsible Party: Sponsor
Other Study IDs: I-009
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2015-09

CONDITIONS: Type II Diabetes
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Manipulation, Chiropractic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chiropractic & Diabetes: All subjects will also receive chiropractic care and receive spinal adjustments as indicated by Basic and Intermediate Activator Methods Protocols, which uses a combination of provocative tests designed to elicit a relative change in leg length in the presence of subluxation. Special shoes designed for improved accuracy of leg length analysis will be used for all visits. The patients will be analyzed two times per week for the first month followed by once per week for the remainder of the study. The Activator Methods protocol will be followed for all visits by all doctors in accordance with the guidelines set forth by Activator Methods International, Ltd. The first four visits will be limited to Basic Protocol to allow the patients to become accustomed to the process.
  Interventions: Other: Chiropractic Adjustment

INTERVENTIONS:
Other: Chiropractic Adjustment — Chiropractic adjustments will be administered using Activator Methods Basic protocol

SUMMARY:
The purpose of this study (15-subject prospective case series) is to examine the effects of the Activator Methods technique on decreasing A1c levels in patients with type II Diabetes Mellitus (aka adult-onset diabetes).

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible to participate in the study if they are between the ages of 30-60 and are clinically diagnosed with Type II diabetes by their primary care providers or endocrinologists (diagnosis usually based on FPG > 126 mg/dL on two occasions).
* Participants must have been diagnosed for at least one year and currently be under medical supervision for the disease.
* They must also have an A1c measurement above 7%, which indicates less than optimal management of the disease.

Exclusion Criteria:

* The study will exclude pregnant women;
* those with co-morbidities affecting life expectancy (e.g. malignancy, CVD); uncontrolled hypertension (> 150/100 mmHg);
* serious trauma (e.g. MVA) within the previous 12 months;
* diagnosed bleeding/clotting disorders; those currently under chiropractic care or having contraindications to Activator care (e.g. vertebral fracture, infection, active inflammatory arthritis, severe osteoporosis).

The presence of these exclusions will be determined during the history and exam procedures. All female subjects will be asked to take precautions during their participation in the study to avoid becoming pregnant.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be eligible to participate in the study if they are between the ages of 30-60 and are clinically diagnosed with Type II diabetes by their primary care providers or endocrinologists (diagnosis usually based on FPG > 126 mg/dL on two occasions). Participants must have been diagnosed for at least one year and currently be under medical supervision for the disease. They must also have an A1c measurement above 7%, which indicates less than optimal management of the disease.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Lowered A1C Levels | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Life University, Marietta, Georgia, United States